CLINICAL TRIAL: NCT03737994
Title: A Biomarker-Driven Protocol for Previously Treated ALK-Positive Non-Squamous NSCLC Patients: The NCI-NRG ALK Protocol
Brief Title: Targeted Treatment for ALK Positive Patients Who Have Previously Been Treated for Non-squamous Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02486; NCI-2018-02486 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU003 (Other: NRG Oncology); NRG-LU003 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — alectinib; brigatinib; Carboplatin; ceritinib; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Crizotinib; ensartinib; lorlatinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- ALK L1198F mutation (alone or combination with ALK inhibitor) (Experimental): Patients with ALK L1198F mutation (alone or in combination with another ALK mutation) receive crizotinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib
- C1156Y (Experimental): Patients with Cy1156Y mutation receive either lorlatinib PO QD, alectinib PO BID, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alectinib; Drug: Brigatinib; Drug: Lorlatinib
- Compound mutation (Experimental): Patients with a compound mutation receive lorlatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lorlatinib
- F1174 (Experimental): Patients with F1174 receive either lorlatinib PO QD, alectinib PO BID, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alectinib; Drug: Brigatinib; Drug: Lorlatinib
- G1202 (including G1202del and G1202R) (Experimental): Patients with G1202 (including G1202del and G1202R) receive either lorlatinib PO QD or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib; Drug: Lorlatinib
- I1171 (Experimental): Patients with I1171 mutation receive either lorlatinib PO QD, ceritinib PO QD, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib; Drug: Ceritinib; Drug: Lorlatinib
- L1196 (including L1196M) (Experimental): Patients with L1196 (including L1196M) mutation receive either lorlatinib PO QD, ceritinib PO QD, alectinib PO BID, brigatinib PO QD, or ensartinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alectinib; Drug: Brigatinib; Drug: Ceritinib; Drug: Crizotinib; Drug: Ensartinib; Drug: Lorlatinib
- MET amplification (Experimental): Patients with MET amplification receive crizotinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib
- No ALK-resistance mutations (Experimental): Patients with no ALK-resistant mutations receive either lorlatinib PO QD, ceritinib PO QD, alectinib PO BID, brigatinib PO QD, ensartinib PO QD, or pemetrexed IV over 10 minutes on day 1 with or without either cisplatin IV or carboplatin IV on day 1. ALK inhibitor cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Pemetrexed-based treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Maintenance treatment of pemetrexed may continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Alectinib; Drug: Brigatinib; Drug: Carboplatin; Drug: Ceritinib; Drug: Cisplatin; Drug: Ensartinib; Drug: Lorlatinib; Drug: Pemetrexed
- V1180 (Experimental): Patients with V1180 mutation receive either lorlatinib PO QD, ceritinib PO QD, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib; Drug: Ceritinib; Drug: Lorlatinib

INTERVENTIONS:
Drug: Alectinib — Given PO
  Other Names: AF 802; AF-802; AF802; Alecensa; ALK Inhibitor RO5424802; CH 5424802; CH-5424802; CH5424802; RG 7853; RG-7853; RG7853; RO 5424802; RO-5424802; RO5424802
  Arms: C1156Y; F1174; L1196 (including L1196M); No ALK-resistance mutations
Drug: Brigatinib — Given PO
  Other Names: Alunbrig; AP 26113; AP-26113; AP26113; Biganib; Briganix; Trepmac
  Arms: C1156Y; F1174; G1202 (including G1202del and G1202R); I1171; L1196 (including L1196M); No ALK-resistance mutations; V1180
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: No ALK-resistance mutations
Drug: Ceritinib — Given PO
  Other Names: LDK 378; LDK-378; LDK378; Zykadia
  Arms: I1171; L1196 (including L1196M); No ALK-resistance mutations; V1180
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: No ALK-resistance mutations
Drug: Crizotinib — Given PO
  Other Names: Alkixen; Crizocent; MET Tyrosine Kinase Inhibitor PF-02341066; PF 02341066; PF-02341066; PF-2341066; PF02341066; Xalkori
  Arms: ALK L1198F mutation (alone or combination with ALK inhibitor); L1196 (including L1196M); MET amplification
Drug: Ensartinib — Given PO
  Other Names: X 396; X-396; X396
  Arms: L1196 (including L1196M); No ALK-resistance mutations
Drug: Lorlatinib — Given PO
  Other Names: 2H-4,8-Methenopyrazolo(4,3-H)(2,5,11)benzoxadiazacyclotetradecine-3-carbonitrile, 7-amino-12-fluoro-10,15,16,17-tetrahydro-2,10,16-trimethyl-15-oxo-, (10R)-; Lorbrena; Lorviqua; PF 06463922; PF-06463922; PF06463922
  Arms: C1156Y; Compound mutation; F1174; G1202 (including G1202del and G1202R); I1171; L1196 (including L1196M); No ALK-resistance mutations; V1180
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: No ALK-resistance mutations

SUMMARY:
This National Cancer Institute (NCI)-NRG ALK Protocol phase II trial studies how well a combination of different biomarker/ALK inhibitors work in treating patients with stage IV ALK positive non-squamous non-small cell lung cancer. Lorlatinib, ceritinib, alectinib, brigatinib, ensartinib, and crizotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as pemetrexed, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether a combination of biomarker/ALK inhibitors or chemotherapy may work better in treating patients with ALK positive non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether ALK kinase domain mutations (G1202/C1156Y/I1171/L1196/ V1180/ F1174/compound mutation) associated with drug resistance are prognostic for objective response to subsequent ALK inhibitor therapy.

II. To assess whether subsequent pemetrexed based chemotherapy improves objective response comparing to ALK inhibitor therapy for no ALK mutation patients.

III. To evaluate objective responses of patients with specific genetic alterations (ALKL1198F/MET double mutation or high-level MET gene amplification) treated with crizotinib.

SECONDARY OBJECTIVES:

I. Progression-free survival (PFS). II. Duration of response (DOR). III. Overall survival (OS). IV. Intracranial objective response rate (ORR). V. Safety and tolerability.

CORRELATIVE SCIENCE OBJECTIVE:

I. Establish concordance between tumor and liquid biopsies.

OUTLINE:

Patients with a G1202R or G1202del mutation receive either lorlatinib orally (PO) once daily (QD) or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a C1156Y mutation receive either lorlatinib PO QD, brigatinib PO QD, or alectinib PO twice daily (BID). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a I1171 mutation receive either lorlatinib PO QD, ceritinib PO QD, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a L1196 mutation receive either lorlatinib PO QD, brigatinib PO QD, ensartinib PO QD, alectinib PO BID, or ceritinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a V1180 mutation receive either lorlatinib PO QD, brigatinib PO QD, or ceritinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a F1174 mutation receive either alectinib PO BID, lorlatinib PO QD, or brigatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with a compound mutation receive lorlatinib PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with an ALK L1198F mutation alone or with another mutation, and patients with high level MET amplification receive crizotinib PO BID. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients with no ALK-resistant mutations receive either lorlatinib PO QD, ceritinib PO QD, alectinib PO BID, brigatinib PO QD, or ensartinib PO QD, or pemetrexed intravenously (IV) over 10 minutes on day 1 and either cisplatin IV or carboplatin IV on day 1. ALK inhibitor cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Pemetrexed-based treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Maintenance treatment of pemetrexed may continue until disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Patients must have histologically or cytologically confirmed stage IV ALK-positive non-squamous non-small cell lung carcinoma (NSCLC) (includes M1a, M1b, M1c stage disease, American Joint Committee on Cancer [AJCC] 8th edition). ALK rearrangement must have been demonstrated by a Food and Drug Administration (FDA) approved assay (Vysis fluorescence in situ hybridization [FISH] or Ventana immunohistochemistry [IHC]) or by next generation sequencing (NGS)
* Patient must be willing and able to undergo a fresh biopsy or if patient has a biopsy after progression on current tyrosine-kinase inhibitor (TKI) within 3 months of study enrollment (and has continued TKI for clinical benefit per treating physician) this tissue may be used. Must have sufficient tissue
* Patient must have progressive disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 after one second generation ALK inhibitor, including LDK378 (ceritinib), alectinib, ensartinib, and brigatinib (may not have received more than one second-generation ALK inhibitor). Patient may have received prior crizotinib; however, the second generation ALK inhibitor received must be the last treatment given prior to study enrollment

  * Prior lorlatinib (third-generation ALK inhibitor) is not allowed
* Prior chemotherapy is not allowed except for one prior cycle received at the time of original diagnosis of metastatic NSCLC with no evidence of disease progression following the cycle. NOTE: prior adjuvant or neoadjuvant chemotherapy is allowed if last dose was received more than 12 months prior to enrollment
* The patient or a legally authorized representative must provide study-specific informed consent prior to Step 1 Registration
* PRIOR TO STEP 2 REGISTRATION
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 (within 28 days prior to step 2 registration)
* Platelets >= 100,000 cells/mm^3 (within 28 days prior to step 2 registration)
* Estimated creatinine clearance >= 60 mL/min by the Cockcroft Gault formula (within 28 days prior to step 2 registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except for patients with documented Gilbert's syndrome) (within 28 days prior to step 2 registration)
* Aspartate aminotransferase (AST) =< 2.5 x ULN; =< 5 x ULN if liver metastases are present (within 28 days prior to step 2 registration)
* Alanine aminotransferase (ALT) =< 2.5 x ULN; =< 5 x ULN if liver metastases are present (within 28 days prior to step 2 registration)
* Patients with asymptomatic treated or untreated brain metastases are eligible. Treated brain metastases are eligible as long as patients have measurable disease outside the brain according to RECIST 1.1. Patients must be on a stable or decreasing dose of steroids for at least 7 days prior to step 2 registration. Anticonvulsants are allowed as long as the patient is neurologically stable and not deteriorating
* Patients enrolled with asymptomatic brain metastases (mets) must have at least one measurable target extracranial lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Acute effects of any prior therapy resolved to baseline severity or to Common Terminology Criteria for Adverse Events (CTCAE) grade =< 1 (except for alopecia, hearing loss)
* Not taking any medications that may interact with selected study medication based on stratification
* Patients must be able to take oral medications (i.e. swallow whole tablets/capsules)
* All females of childbearing potential must have a blood test or urine study within 14 days prior to Step 2 Registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
  * Women must not be pregnant or breast-feeding due to potential harm to the fetus or infant from ALK inhibitors and the unknown risk. Women of childbearing potential and sexually active males must agree to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study

Exclusion Criteria:

* Major surgery within 2 weeks of study entry. Minor surgical procedures (e.g., port insertion, pleurex catheter placement) are allowed and all wounds must not show signs of infection or draining
* Palliative RT (< 10 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have completed at least 1 week prior to study entry. Whole brain RT or other palliative RT must have been completed at least 2 weeks prior to study entry
* Prior dose of next generation ALK inhibitor (LDK378 [ceritinib], alectinib, ensartinib, lorlatinib) within 5 days prior to step 2 registration. Prior dose of brigatinib within 7 days prior to step 2 registration
* History of interstitial lung disease or interstitial fibrosis, including a history of pneumonitis, obliterative bronchiolitis, pulmonary fibrosis. Patients with a history of prior radiation pneumonitis are not excluded
* Active inflammatory gastrointestinal disease (such as Crohns, ulcerative colitis), chronic diarrhea, symptomatic diverticular disease, or any gastrointestinal disease that would affect the absorption of oral medications or increase the risk of toxicity
* Clinically significant cardiovascular abnormalities, as determined by the treating/registering physician, such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia, or myocardial infarction within 6 months
* Active and clinically significant bacterial, fungal, or viral infection
* Patients with active or chronic pancreatitis based on lipase elevation, symptoms, and radiographic findings
* Other concomitant serious illness or organ system dysfunction that in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the study drug
* Patients must not plan to receive any other investigational agents during the course of therapy
* Patients with active malignancy other than ALK-positive non-squamous NSCLC within the last 2 years are excluded (note: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, papillary thyroid cancer treated with curative intent, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for 2 years are eligible)
* No chemotherapy and/or immunotherapy allowed after step 1 registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2025-12-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Lin, Principal Investigator — NRG Oncology
Locations (491):
- United States (491):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - 21st Century Oncology - El Segundo, El Segundo, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - GenesisCare USA - Boca Raton FP02, Boca Raton, Florida
  - GenesisCare USA - Boca Ration FP06, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - GenesisCare USA - Key West, Key West, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - GenesisCare USA - Palm Beach Gardens, Palm Beach Gardens, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Cancer Center-Bethel Park, Bethel Park, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Oncology Hematology Association, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Saint Clair Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Tissue and blood submissions were required after first step registration, before second step registration (treatment assignment). Of 16 participants screened, 10 were assigned to treatment.
Groups:
- Lorlatinib: Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations, compound mutation*, or no mutations, can be assigned to receive lorlatinib. *Compound mutation = two or more resistance mutation excluding those with L1198F or L1189F/MET amplification = L1198F mutation alone or in combination, or no anaplastic lymphoma kinase (ALK) mutation but any MET amplification.
  Lorlatinib: 100 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- LDK378 (Ceritinib): Participants with I1171, L1196 (including L1196M), or V1180 mutations, or no having no ALK-resistance mutations or MET amplifications, can be assigned to receive ceritinib
  Ceritinib: 450 mg orally once a day with food. Treatment continues until disease progression or unacceptable toxicity.
- Alectinib: Participants with C1156Y, L1196 (including L1196M), or F1174 mutations, or no having no ALK-resistance mutations or MET amplifications, can be assigned to receive Alectinib.
  Alectinib: 600 mg orally twice daily with food. Treatment continues until disease progression or unacceptable toxicity.
- Brigatinib: Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations, or having no ALK-resistance mutations or MET amplifications, can be assigned to receive brigatinib.
  Brigatinib: 90 mg orally once a day (with or without food) for the first 7 days; if tolerated, with no respiratory symptoms, increase the dose to 180 mg once daily. Treatment continues until disease progression or unacceptable toxicity.
- Ensartinib: Participants with L1196 (including L1196M) mutations or having no ALK-resistance mutations or MET amplifications can be assigned to receive ensartinib.
  Ensartinib: 225 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- Crizotinib: Participants with ALK L1198F (alone/ in combination with another ALK mutation) or mesenchymal-to-epithelial transition (MET) amplification can be assigned to receive crizotinib
  Crizotinib: 250 mg orally twice daily with or without food. Treatment continues until disease progression or unacceptable toxicity.
- Pemetrexed +/- Cisplatin or Carboplatin: Participants with no ALK-resistance mutations or MET amplifications can be assigned to receive pemetrexed, which optionally can be combined with cisplatin or carboplatin.
  Carboplatin: Carboplatin is optional. Dosing of area under the curve (AUC) = 5 once every 3 weeks (on Day 1 of a 21 day cycle with pemetrexed) intravenously, prepared and administered per institution policy. Continues for 4-6 cycles.
  Cisplatin: Cisplatin is optional. 75 mg/m^2 intravenously once every 3 weeks (on Day 1 of a 21 day cycle with pemetrexed), prepared and administered per institution policy.
  Pemetrexed: Pemetrexed may be given alone or with either cisplatin or carboplatin. Pemetrexed 500 mg/m2 administered intravenously on Day 1 of a 21 day cycle, optionally with cisplatin or carboplatin for 4-6 cycles. Then pemetrexed (as a single agent) continues until progression or significant toxicity.
Period: Overall Study
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Alectinib | Brigatinib | Ensartinib | Crizotinib | Pemetrexed +/- Cisplatin or Carboplatin
Started | 3 | 1 | 0 | 2 | 3 | 0 | 1
Disease Assessment Population (Eligible participants who started protocol treatment and had post-baseline disease assessment.) | 3 | 1 | 0 | 2 | 2 | 0 | 0
Survival Population (Eligible participants who started protocol treatment and have post-baseline survival status.) | 3 | 1 | 0 | 2 | 3 | 0 | 0
Adverse Event Population (Eligible participants who started protocol treatment and have adverse event data.) | 3 | 1 | 0 | 2 | 3 | 0 | 0
Completed (Participants contributing data to any results are considered to have completed the study.) | 3 | 1 | 0 | 2 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants assigned to treatment (second step registration)
Groups:
- Lorlatinib: Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations, compound mutation*, or no mutations, can be assigned to receive lorlatinib. *Compound mutation = two or more resistance mutation excluding those with L1198F or L1189F/MET amplification = L1198F mutation alone or in combination, or no ALK mutation but any MET amplification.
  Lorlatinib: 100 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Brigatinib | Ensartinib | Pemetrexed +/- Cisplatin or Carboplatin | Total
Number analyzed (Participants) | 3 | 1 | 2 | 3 | 1 | 10
Age, Customized [Count of Participants; unit: Participants]
  <= 49 years | 1 | 1 | 2 | 1 | 0 | 5
  50-59 years | 1 | 0 | 0 | 1 | 0 | 2
  60-69 years | 1 | 0 | 0 | 1 | 0 | 2
  >= 70 years | 0 | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 1 | 7
  Male | 1 | 1 | 0 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 1 | 1 | 3 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 3 | 0 | 2 | 3 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Mutation [Count of Participants; unit: Participants]
  I1171 | 1 | 1 | 1 | 0 | 0 | 3
  No ALK-resistance mutation / MET amplification | 2 | 0 | 1 | 3 | 1 | 7
Has CNS metastases [Count of Participants; unit: Participants] | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Per Investigator Assessment Using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria
Description: ORR= number of subjects with best overall response (BOR) of complete or partial response (CR, PR) divided by number of evaluable subjects. BOR= best response recorded from start of treatment to first progression (PD)/new anticancer therapy, otherwise last follow-up.
  * CR: disappearance of target and non-target lesions; no new lesions; pathological lymph nodes < 10mm.
  * PR: 30% decrease in target lesions; non-target lesions not progressed or not evaluated; no new lesions.
  * PD: 20% increase of target lesions and/or new lesion(s).
  ORR was to be compared using Fisher's exact test within each ALK inhibitor treatment arm (each mutation vs. no mutation) and also within the subset of subjects with no mutation comparing each experimental arm vs. pemetrexed. Due to early accrual closure (few subjects), only the number of subjects with BOR of CR or PR are provided, by mutation, no statistical testing. Analysis was to occur after each patient was potentially followed ≥ 24 weeks.
Time Frame: Baseline to 24 weeks
Population: Eligible participants who started protocol treatment and had post-baseline disease assessment. Treatment arms with no evaluable participants are not shown.
Measure: Count of Participants; unit: Participants
Groups:
- Lorlatinib: Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations, compound mutation*, or having no ALK-resistance mutations or MET amplifications, can be assigned to receive lorlatinib. *Compound mutation = two or more resistance mutation excluding those with L1198F or L1189F/MET amplification = L1198F mutation alone or in combination, or no ALK mutation but any MET amplification.
  Lorlatinib: 100 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- LDK378 (Ceritinib): Participants with I1171, L1196 (including L1196M), or V1180 mutations, or no having no ALK-resistance mutations or MET amplifications, can be assigned to receive ceritinib.
  Ceritinib: 450 mg orally once a day with food. Treatment continues until disease progression or unacceptable toxicity.
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Brigatinib | Ensartinib
Number analyzed (Participants) | 3 | 1 | 2 | 2
Participants
  Mutation = I1171: BOR of CR or PR: number analyzed (Participants) | 1 | 1 | 1 | 0
  Mutation = I1171: BOR of CR or PR | 1 | 0 | 0 |
  Mutation = None: BOR of CR or PR: number analyzed (Participants) | 2 | 0 | 1 | 2
  Mutation = None: BOR of CR or PR | 2 |  | 1 | 0

2. Secondary Outcome: Progression-free Survival (PFS), Per Investigator Assessment Using RECIST v1.1 Criteria
Description: Progression-free survival time is defined as the time from second step registration to the date of the first disease progression / progressive disease (PD), death, or last known follow-up (censored). Progressive disease is defined as a 20% increase of target lesions and/or new lesion(s). Percentage of participants progression-free at a given time (PFS) was to be estimated by the Kaplan-Meier method. Median PFS and PFS at specific time points was to be reported, with 95% confidence intervals, for each mutation (or no mutation)/regimen combination. Due to early accrual closure resulting in few participants, only the number of participants who progressed or died, by mutation, with no statistical testing.
Time Frame: Baseline to the date of the first disease progression / progressive disease, death, or last known follow-up. Maximum follow-up time was 33.6 months, median 8.9 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Brigatinib | Ensartinib
Number analyzed (Participants) | 3 | 1 | 2 | 2
Participants
  Mutation = I1107: progression or death: number analyzed (Participants) | 1 | 1 | 1 | 0
  Mutation = I1107: progression or death | 0 | 0 | 1 |
  Mutation = none: progression or death: number analyzed (Participants) | 2 | 0 | 1 | 2
  Mutation = none: progression or death | 1 |  | 1 | 2

3. Secondary Outcome: Duration of Overall Response, Per Investigator Assessment Using RECIST v1.1
Description: Duration of overall response (DOR) is defined as the time from the first occurrence of a documented BOR of CR or PR to the first date of recorded disease progression (PD) or death from any cause (whichever occurs first). BOR is the best response recorded from the start of treatment to first progression (PD)/new anticancer therapy, otherwise last follow-up.
  * CR: disappearance of target and non-target lesions; no new lesions; pathological lymph nodes < 10mm.
  * PR: 30% decrease in target lesions; non-target lesions not progressed or not evaluated; no new lesions.
  * PD: 20% increase of target lesions and/or new lesion(s).
  Median DOR was to be estimated, with 95% confidence intervals, for each mutation/regimen combination using the Kaplan-Meier method. Due to early accrual closure resulting in few subjects, only the mean and range DOR are provided, by mutation, and no statistical testing was done.
Time Frame: as for outcome 2
Population: Eligible participants who started protocol treatment and had complete or partial response. Treatment arms with no evaluable participants are not shown.
Measure: Mean (Full Range); unit: months
Arm/Group | Lorlatinib | Brigatinib
Number analyzed (Participants) | 3 | 1
months
  Mutation = I1171: number analyzed (Participants) | 1 | 0
  Mutation = I1171 | 27.9 [27.9 to 27.9] |
  Mutation = None: number analyzed (Participants) | 2 | 1
  Mutation = None | 19.2 [9.4 to 29.1] | 3.5 [3.5 to 3.5]

4. Secondary Outcome: Overall Survival (OS)
Description: Survival time is defined as the time from second step registration to the date of death, or last known follow-up (censored). Percentage of participants alive at a given time (OS) was to be estimated by the Kaplan-Meier method. Median OS and OS at specific time points was to be reported, with 95% confidence intervals, for each mutation/regimen combination. Due to early accrual closure resulting in few patients, only the number of participants who died are provided, by mutation, and no statistical testing was done.
Time Frame: Baseline to the date of death or last known follow-up. Maximum follow-up time was 33.6 months, median 8.9 months.
Population: Eligible participants who started protocol treatment, with post-baseline survival status. Treatment arms with no evaluable participants are not shown.
Measure: Count of Participants; unit: Participants
Groups:
- LDK378 (Ceritinib): Participants with I1171, L1196 (including L1196M), or V1180 mutations, or having no ALK-resistance mutations or MET amplifications, can be assigned to receive ceritinib
  Ceritinib: 450 mg orally once a day with food. Treatment continues until disease progression or unacceptable toxicity.
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Brigatinib | Ensartinib
Number analyzed (Participants) | 3 | 1 | 2 | 3
Participants
  Mutation = I1171: deaths: number analyzed (Participants) | 1 | 1 | 1 | 0
  Mutation = I1171: deaths | 0 | 0 | 0 |
  Mutation = None: deaths: number analyzed (Participants) | 2 | 0 | 1 | 3
  Mutation = None: deaths | 0 |  | 1 | 2

5. Secondary Outcome: Intracranial Objective Response Rate, Per Investigator Assessment Using RECIST v1.1
Description: Intracranial objective response rate (IORR) is defined as the number of participants with central nervous system (CNS) metastasis complete or partial response (CR, PR) divided by the number of evaluable participants with baseline CNS metastasis and no prior CNS radiation therapy. Participants who required additional treatment (for their non-cranial systemic disease) would be considered as non-responders (if they have not previously had an intracranial response).
  * CR: disappearance of target and non-target lesions; no new lesions; pathological lymph nodes < 10mm.
  * PR: 30% decrease in target lesions; non-target lesions not progressed or not evaluated; no new lesions.
  IORR was to be estimated for each mutation/regimen combination, with the associated 95% confidence intervals (using Clapper-Pearson method). Due to early accrual closure resulting in few subjects, only the number of subjects with CR or PR are provided, by mutation, with no statistical testing.
Time Frame: Baseline to 24 weeks
Population: No participants with baseline CNS metastasis had evaluable post-baseline CNS metastasis assessment.
Arm/Group | Lorlatinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: Baseline to the date of last known follow-up. Maximum follow-up time was 33.6 months, median 8.9 months.
Population: Eligible participants who started protocol treatment, with adverse event data. Treatment arms with no evaluable participants are not shown.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Brigatinib | Ensartinib
Number analyzed (Participants) | 3 | 1 | 2 | 3
Participants
  Mutation = I1107: number analyzed (Participants) | 1 | 1 | 1 | 0
  Mutation = I1107: Grade 1 | 0 | 0 | 0 |
  Mutation = I1107: Grade 2 | 0 | 0 | 0 |
  Mutation = I1107: Grade 3 | 1 | 1 | 1 |
  Mutation = I1107: Grade 4 | 0 | 0 | 0 |
  Mutation = I1107: Grade 5 | 0 | 0 | 0 |
  Mutation = none: number analyzed (Participants) | 2 | 0 | 1 | 3
  Mutation = none: Grade 1 | 0 |  | 0 | 0
  Mutation = none: Grade 2 | 0 |  | 0 | 0
  Mutation = none: Grade 3 | 2 |  | 0 | 3
  Mutation = none: Grade 4 | 0 |  | 0 | 0
  Mutation = none: Grade 5 | 0 |  | 1 | 0

7. Other Pre Specified Outcome: Agreement of Biopsy Mutation and Circulating Free Deoxyribonucleic Acid (cfDNA) Mutation Results
Description: For each mutation, the agreement of the biopsy result (present, absent, unavailable) and the cfDNA result (present, absent, unavailable) would be assessed. Agreement of cfDNA and biopsy results will be considered separately for MET amplification and for the gene mutations. This outcome measure was to be contingent upon FDA approval of the outcome measure analysis plan, which was not pursued due to the early accrual closure.
Time Frame: Baseline
Population: No assay data for analysis was received.
Groups:
- LDK378 (Ceritinib): Participants with I1171, L1196 (including L1196M), or V1180 mutations, or having no having no ALK-resistance mutations or MET amplifications, can be assigned to receive ceritinib
  Ceritinib: 450 mg orally once a day with food. Treatment continues until disease progression or unacceptable toxicity.
- Alectinib: Participants with C1156Y, L1196 (including L1196M), or F1174 mutations, or having no ALK-resistance mutations or MET amplifications, can be assigned to receive Alectinib.
  Alectinib: 600 mg orally twice daily with food. Treatment continues until disease progression or unacceptable toxicity.
Arm/Group | Lorlatinib | LDK378 (Ceritinib) | Alectinib | Brigatinib | Ensartinib | Crizotinib | Pemetrexed +/- Cisplatin or Carboplatin
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to the date of last known follow-up. Maximum follow-up time was 33.6 months, median 8.9 months.
Description: Note, treatment arms are reported by mutation / no mutation.
Groups:
- Lorlatinib (Mutations): Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations, or compound mutation*. *Compound mutation = two or more resistance mutation excluding those with L1198F or L1189F/MET amplification = L1198F mutation alone or in combination, or no ALK mutation but any MET amplification.
  Lorlatinib: 100 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- Lorlatinib (no Mutations): Participants with no ALK-resistance mutations or MET amplifications.
  Lorlatinib: 100 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
- LDK378 (Ceritinib): Participants with I1171, L1196 (including L1196M), or V1180 mutations.
  Ceritinib: 450 mg orally once a day with food. Treatment continues until disease progression or unacceptable toxicity.
- Brigatinib (Mutations): Participants with G1202 (including G1202del and G1202R), C1156Y, I1171, L1196 (including L1196M), V1180, or F1174 mutations.
  Brigatinib: 90 mg orally once a day (with or without food) for the first 7 days; if tolerated, with no respiratory symptoms, increase the dose to 180 mg once daily. Treatment continues until disease progression or unacceptable toxicity.
- Brigatinib (no Mutations): Participants with no ALK-resistance mutations or MET amplifications.
  Brigatinib: 90 mg orally once a day (with or without food) for the first 7 days; if tolerated, with no respiratory symptoms, increase the dose to 180 mg once daily. Treatment continues until disease progression or unacceptable toxicity.
- Ensartinib: Participants with no ALK-resistance mutations or MET amplifications.
  Ensartinib: 225 mg orally once a day with or without food. Treatment continues until disease progression or unacceptable toxicity.
Arm/Group | Lorlatinib (Mutations) | Lorlatinib (no Mutations) | LDK378 (Ceritinib) | Brigatinib (Mutations) | Brigatinib (no Mutations) | Ensartinib
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/1 | 1/1 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 0/1 | 0/1 | 1/1 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/1 | 1/1 | 1/1 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (Mutations) (N=1) | Lorlatinib (no Mutations) (N=2) | LDK378 (Ceritinib) (N=1) | Brigatinib (Mutations) (N=1) | Brigatinib (no Mutations) (N=1) | Ensartinib (N=3)
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib (Mutations) (N=1) | Lorlatinib (no Mutations) (N=2) | LDK378 (Ceritinib) (N=1) | Brigatinib (Mutations) (N=1) | Brigatinib (no Mutations) (N=1) | Ensartinib (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0 | 2
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalized edema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cholesterol high (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Serum amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 10 subjects randomized out of 660 planned. Study assessments and data collection continued only for those participants still receiving study treatment and ceased at treatment completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval from the sponsor. In addition, PI's are required to abide by Collaborator's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03737994/Prot_SAP_000.pdf
  • Informed Consent Form: Treatment with Alectinib (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03737994/ICF_001.pdf
  • Informed Consent Form: Treatment with Brigatinib (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03737994/ICF_002.pdf
  • Informed Consent Form: Treatment with LDK378 (Ceritinib) (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03737994/ICF_003.pdf